CLINICAL TRIAL: NCT04243993
Title: Clinical Outcomes of Bio-MA and ProRoot MTA in Non-surgical and Surgical Endodontic Treatment: a Randomized Controlled Clinical Trial
Brief Title: Clinical Outcomes of Bio-MA and ProRoot MTA in Endodontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-DT/PY-IRB 2016/052.0310
Record Dates: First submitted 2019-12-24; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Clinical Outcome; Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-MA (Other): Calcium silicate cement containing calcium chloride accelerator
  Interventions: Other: Calcium silicate cement
- ProRoot MTA (Other): Calcium silicate cement without calcium chloride accelerator
  Interventions: Other: Calcium silicate cement

INTERVENTIONS:
Other: Calcium silicate cement — Calcium silicate cement for using in endodontic treatments i.e. pulpotomy, orthograde MTA apical barrier, root perforation repair, and endodontic microsurgery.

SUMMARY:
The purpose of this study is to compare the endodontic outcomes of Bio-MA and ProRoot MTA in pulpotomy, orthograde MTA apical barrier, root perforation repair, endodontic microsurgery.

DETAILED DESCRIPTION:
The patients were recruited at the Endodontic clinic, Faculty of Dentistry, Mahidol University, Thailand. Each treatment was provided following the standard protocol. The calcium silicate based material (Bio-MA or ProRoot MTA) was randomly selected and used in the treatment. The patients were periodically recalled at 6 to 12 months. The outcome of the three treatments based on the clinical and radiographic criteria was assessed by the calibrated examiners and interpreted as ''healed/healing" or ''disease.''

ELIGIBILITY:
Inclusion Criteria:

* Teeth treated with pulpotomy, orthograde MTA apical barrier, root perforation repair or endodontic microsurgery

Exclusion Criteria:

* Teeth with un-restorable condition
* Teeth with crack or fracture
* Teeth with external or internal root resorption
* Teeth with chronic periodontitis with marginal bone loss more than 5 mm

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Healed rate | At least 1 year recall
  No clinical sign and symptoms and periapical area in radiograph is normal. Describe in percentage.
Healing rate | At least 1 year recall
  No clinical sign and symptoms and periapical lesion in radiograph is reduce in size. Describe in percentage.
Disease rate | At least 1 year recall
  Clinical sign and symptoms is present and/or periapical lesion in radiograph is unchange or enlarge. Describe in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Supachai Sutimuntanakul, TBOD, Study Director — Mahidol University
Locations (1):
- Nuttida Tungsuksomboon, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No